CLINICAL TRIAL: NCT01773382
Title: The Effects of Weight Reduction in Chronic Proteinuric IgA Nephropathy
Brief Title: The Effects of Weight Reduction in IgA Nephropathy
Acronym: WeightPro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Talerngsak Kanjanabuch, Kidney and metabolic research center, Faculty of medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PK8197
Record Dates: First submitted 2013-01-04; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Proteinuria
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): standard treatment of IgA nephropathy including ACEI/ARB for blood pressure control (target BP <130/80 mmHg)
- weight reduction (Experimental): target weight reduction is 3-5% from baseline
  Interventions: Behavioral: weight reduction

INTERVENTIONS:
Behavioral: weight reduction — 1. Set target daily energy requirement by nutritionist (25-30 Kcal/Kg/day minus 500 Kcal)
  2. Advice and encourage patients to do aerobic exercise at least 30 minutes/day for 4-5 days/weeks.
  3. Daily body weight measurement.
  4. Record food diary
  Other Names: controlled weight reduction program
  Arms: weight reduction

SUMMARY:
The study aims to explore the non-pharmacological treatment of IgA nephropathy by weight reduction. The investigators hypothesized that benefits of weight loss may reduce proteinuria.

DETAILED DESCRIPTION:
This is a prospective randomized study in adult IgA nephropathy. The investigators enrolled 30 patients who have proteinuria exceeds 1 g per day with biopsy proven IgA nephropathy. The experimental arm recieves the non-pharmacological treatment, weight reduction protocol. All patients in this arm must be reduce their body weight in 3-5 % from baseline as protocol. Another arm is control group which recieves standard treatment of IgA nephropathy including ACEIs/ARBs for blood pressure control (target < 130/80 mmHg). The primary outcome is proteinuria level. The secondary outcome is cytokines and inflammatory markers level including interleukin-6, resistin, adiponectin, leptin and monocyte chemoattractant protein-1.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven IgA nephropathy
* body mass index more than 23 Kg/m2
* 24 hours urine protein more than 1 g
* estimated GFR more than 20 ml/min

Exclusion Criteria:

* pregnancy and lactation
* rapidly renal function decline
* crescent formation in renal biopsy more than 10%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Percentage change of 24-hour proteinuria | 6 months
  The investigators measure amount of 24-hour proteinuria at randomization peroid ( as baseline), first, third and sixth month. Then, investigators calculate the percentage reduction of proteinuria at different time points.

SECONDARY OUTCOMES:
plasma concentration of IL-6, adiponectin, resistin, leptin, MCP-1 | 6 months
  The investigators measure amount of plasma concentration of IL-6, adiponectin, resistin, leptin, MCP-1 at randomization peroid ( as baseline) and sixth month. Then, investigators calculate the percentage reduction of these cytokines in 6 months peroid.

CONTACTS AND LOCATIONS:
Overall Officials: Piyawan Kittiskulnam, M.D., Study Director — Chulalongkorn University
Locations (1):
- Faculty of medicine, Chulalongkorn university, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940